CLINICAL TRIAL: NCT03755518
Title: A Phase 3b, Multicenter, Single-Arm, Open-Label Efficacy and Safety Study of Fedratinib in Subjects With DIPSS (Dynamic International Prognostic Scoring System)-Intermediate or High-Risk Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (Post-PV MF), or Post-Essential Thrombocythemia Myelofibrosis (Post-ET MF) and Previously Treated With Ruxolitinib
Brief Title: A Trial of Fedratinib in Subjects With DIPSS, Intermediate or High-Risk Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocythemia Myelofibrosis and Previously Treated With Ruxolitinib
Acronym: FREEDOM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Celgene (Industry)
Collaborators: Impact Biomedicines, Inc., a wholly owned subsidiary of Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEDR-MF-001; U1111-1223-2862 (Other: WHO); 2018-002237-38 (EudraCT Number)
Expanded Access: NCT03723148 (Available)
Record Dates: First submitted 2018-11-08; First posted 2018-11-28 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: Myelofibrosis (MF); Primary Myelofibrosis (PMF); Post-Polycythemia Vera Myelofibrosis (Post-PV); Post-essential thrombocythemia Myelofibrosis (Post-ET); Myeloproliferative neoplasms (MPN)
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of Fedratinib 400mg/day (Experimental): Self-administered Investigational Product (IP) (400 mg/day) on an outpatient basis, once daily preferably with food during an evening meal at the same time each day in consecutive 4-week (28-day) cycles.
  Interventions: Drug: FEDRATINIB

INTERVENTIONS:
Drug: FEDRATINIB — A potent and selective inhibitor of JAK2 kinase activity

SUMMARY:
This is Single-Arm, Open-Label Efficacy and Safety Trial of Fedratinib in Subjects with DIPSS (Dynamic International Prognostic Scoring System)-Intermediate or High- Risk Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (post-PV MF), or Post-Essential Thrombocythemia Myelofibrosis (post-ET MF) and Previously Treated with Ruxolitinib.

The primary objective of the study is to evaluate the percentage of subjects with at least a 35% reduction in spleen size and one of the secondary objectives is to evaluate the safety of fedratinib.

DETAILED DESCRIPTION:
This is Single-Arm, Open-Label Efficacy and Safety Trial of Fedratinib in Subjects with DIPSS (Dynamic International Prognostic Scoring System)-Intermediate or High- Risk Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (post-PV MF), or Post-Essential Thrombocythemia Myelofibrosis (post-ET MF) and Previously Treated with Ruxolitinib.

The spleen volume reduction at the end of Cycle 6 as the primary objective. The secondary objectives of the study are to further evaluate the safety and to assess and implement mitigation strategies for WE and for gastrointestinal (GI) adverse events.

The study will be at multiple centers to provide access to a broad population and have assurance the results are likely to have general applicability.

This is also conducted as an open-label study to collect efficacy and safety data with fedratinib use, no randomization or stratification will occur.

ELIGIBILITY:
Inclusion Criteria:

Main Study Inclusion Criteria

1. Subject is at least 18 years of age at the time of signing the informed consent form (ICF)
2. Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) of 0, 1 or 2
3. Subject has diagnosis of primary myelofibrosis (PMF) according to the 2016 World Health Organization (WHO) criteria, or diagnosis of post-ET or post-PV myelofibrosis according to the IWG-MRT 2007 criteria, confirmed by the most recent local pathology report
4. Subject has a DIPSS Risk score of Intermediate or High
5. Subject has a measurable splenomegaly during the screening period as demonstrated by spleen volume of ≥ 450 cm3 by MRI or CT-scan assessment or by palpable spleen measuring ≥ 5 cm below the left costal margin.
6. Subject has been previously exposed to ruxolitinib, while diagnosed with MF (PMF, post-ET MF or post-PV MF), and must meet at least one of the following criteria (a or b)

   1. Treatment with ruxolitinib for ≥ 3 months
   2. Treatment with ruxolitinib for ≥ 28 days complicated by any of the following:

      * Development of a red blood cell transfusion requirement (at least 2 units/month for 2 months) or
      * Grade ≥ 3 AEs of thrombocytopenia, anemia, hematoma, and/or hemorrhage while on treatment with ruxolitinib
7. Subject must have treatment-related toxicities from prior therapy resolved to Grade 1 or pretreatment baseline before start of last therapy prior to fedratinib treatment.
8. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted
9. Subject is willing and able to adhere to the study visit schedule and other protocol requirements
10. Participants must agree to use effective contraception

Exclusion Criteria:

Main Study Exclusion Criteria

1. Any of the following laboratory abnormalities:

   1. Platelets < 50,000/μL
   2. Absolute neutrophil count (ANC) < 1.0 x 109/L
   3. White blood count (WBC) > 100 x 10^9/L
   4. Myeloblasts > 5 % in peripheral blood
   5. Estimated glomerular filtration rate < 30 mL/min/1.73 m^2 (as per the Modification of Diet in Renal Disease [MDRD] formula)
   6. Serum amylase or lipase > 1.5 x ULN (upper limit of normal)
   7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x ULN
   8. Total bilirubin > 1.5 x ULN, subject's total bilirubin between 1.5 - 3.0 x ULN are eligible if the direct bilirubin fraction is < 25% of the total bilirubin
2. Subject is pregnant or lactating female
3. Subject with previous splenectomy
4. Subject with previous or planned hematopoietic cell transplant
5. Subject with prior history of encephalopathy, including Wernicke's
6. Subject with signs or symptoms of encephalopathy including Wernicke's (eg, severe ataxia, ocular paralysis or cerebellar signs)
7. Subject with thiamine deficiency, defined as thiamine levels in whole blood below normal range according to institutional standard and not corrected prior to enrollment on the study
8. Subject with concomitant treatment with or use of pharmaceutical, herbal agents or food known to be strong or moderate inducers of Cytochrome P450 3A4 (CYP3A4), or dual CYP2C19 and CYP3A4 inhibitors
9. Subject on any chemotherapy, immunomodulatory drug therapy (eg, thalidomide, interferon-alpha), anagrelide, immunosuppressive therapy, systemic corticosteroids > 10 mg/day prednisone or equivalent. Subjects who have had prior exposure to hydroxyurea (eg, Hydrea) in the past may be enrolled into the study as long as it has not been administered within 14 days prior to the start of fedratinib treatment
10. Subject has received ruxolitinib within 14 days prior to the start of fedratinib
11. Subject on treatment with myeloid growth factor (eg, granulocyte-colony stimulating factor [G-CSF]) within 14 days prior to the start of fedratinib treatment
12. Subject with previous exposure to Janus kinase (JAK) inhibitor(s) for more than 1 cycle other than ruxolitinib treatment
13. Subject on treatment with aspirin with doses > 150 mg daily
14. Subject with major surgery within 28 days before starting fedratinib treatment
15. Subject with diagnosis of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemochromatosis, non-alcoholic steatohepatitis)
16. Subject with prior malignancy other than the disease under study unless the subject has not required treatment for the malignancy for at least 3 years prior to enrollment.

    However, subject with the following history/concurrent conditions provided successfully treated may enroll: non-invasive skin cancer, in situ cervical cancer, carcinoma in situ of the breast, incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system), or is free of disease and on hormonal treatment only
17. Subject with uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4)
18. Subject with known human immunodeficiency virus (HIV), known active infectious Hepatitis B (HepB), and/or known active infectious Hepatitis C (HepC)
19. Subject with serious active infection
20. Subject with presence of any significant gastric or other disorder that would inhibit absorption of oral medication
21. Subject is unable to swallow capsule
22. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
23. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
24. Subject has any condition that confounds the ability to interpret data from the study
25. Subject with participation in any study of an investigational agent (drug, biologic, device) within 30 days prior to start of fedratinib treatment
26. Subject with life expectancy of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (28):
  - Local Institution - 117, Aurora, Colorado
  - Local Institution - 126, Miami, Florida
  - Local Institution - 113, Augusta, Georgia
  - Local Institution - 112, Chicago, Illinois
  - Local Institution - 109, Chicago, Illinois
  - Local Institution - 121, Park Ridge, Illinois
  - Local Institution - 100, Kansas City, Kansas
  - Local Institution - 123, Baltimore, Maryland
  - Local Institution - 118, Bethesda, Maryland
  - Local Institution - 127, Columbia, Maryland
  - Local Institution - 103, Ann Arbor, Michigan
  - Local Institution - 101, St Louis, Missouri
  - Local Institution - 128, Newark, New Jersey
  - Local Institution - 130, Brooklyn, New York
  - Local Institution - 115, New York, New York
  - Local Institution - 124, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Local Institution - 105, Chapel Hill, North Carolina
  - Local Institution - 114, Durham, North Carolina
  - Local Institution - 111, Cincinnati, Ohio
  - Local Institution - 106, Pittsburgh, Pennsylvania
  - Local Institution - 108, Sioux Falls, South Dakota
  - Local Institution - 119, Dallas, Texas
  - Local Institution - 132, Fort Worth, Texas
  - Local Institution - 110, Houston, Texas
  - Local Institution - 120, San Antonio, Texas
  - Local Institution - 116, Seattle, Washington
  - Local Institution - 129, Madison, Wisconsin
- Canada (7):
  - Local Institution - 203, Vancouver, British Columbia
  - Local Institution - 207, London, Ontario
  - Local Institution - 205, Ottawa, Ontario
  - Local Institution - 200, Toronto, Ontario
  - Local Institution - 201, Montreal, Quebec
  - Local Institution - 202, Montreal, Quebec
  - Local Institution - 204, Sherbrooke, Quebec

REFERENCES:
- [Derived] Gupta V, Yacoub A, Mesa RA, Harrison CN, Vannucchi AM, Kiladjian JJ, Deeg HJ, Fazal S, Foltz L, Mattison RJ, Miller CB, Parameswaran V, Brown P, Hernandez C, Wang J, Talpaz M. Safety and efficacy of fedratinib in patients with myelofibrosis previously treated with ruxolitinib: primary analysis of FREEDOM trial. Leuk Lymphoma. 2024 Sep;65(9):1314-1324. doi: 10.1080/10428194.2024.2346733. Epub 2024 Jun 5. PMID 38838026
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Fedratimib: 400 mg/day PO (4 x 100 mg capsules)
Period: Overall Study
Arm/Group | Fedratimib
Started | 38
Completed (Completed = continuing treatment) | 0
Not Completed | 38
Not completed — Lack of Efficacy | 10
Not completed — Adverse Event | 7
Not completed — Study Terminated by Sponsor | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Progressive Disease | 4
Not completed — Bone Marrow Transplant | 4
Not completed — Physicians Decision | 1
Not completed — Relapse | 1
Not completed — Withdrawal by Investigator for Non Compliance | 1
Not completed — Withdrawal by PI | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
EE Population [Number; unit: Participants] — Efficacy Evaluable Population
  All participants who enrolled and received at least one dose of fedratinib, had an evaluable spleen volume at baseline (based on MRI/CT scan) and at least one post-baseline response assessment by MRI/CT scan
  Participants | 35
MFSAF Population [Number; unit: Participants] — fedratinib treated participants with a Total Symptom Score (TSS) at baseline (eg, symptom score) > 0 and at least 1 post baseline TSS assessment
  Participants | 36
Palpation evaluable population [Number; unit: Participants] — All participants who enrolled and received at least one dose of fedratinib, and had an enlarged spleen ≥ 5 cm below LCM at baseline
  Participants | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have a ≥ 35% Spleen Volume Reduction (SVR) at End of Cycle 6
Description: Percentage of participants who have a ≥ 35% SVR at end of Cycle 6 as compared to baseline. Participants with a missing MRI/CT spleen volume at the end of Cycle 6 including those who meet the criteria for progression of splenomegaly before the end of Cycle 6 will be considered non-responders. Baseline value is defined as the last value or measurement taken prior to the first dose in the study
Time Frame: From First Dose to end of Cycle 6 (approximately 168 days)
Population: Efficacy evaluable population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 35
Percentage of participants | 25.7 [12.5 to 43.3]

2. Secondary Outcome: Number of Participants of All Grade Adverse Events (AEs) and Grade 3/4 AEs
Description: Number of participants and severity of all grade adverse events (AEs) and grade 3/4 AEs as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.
Time Frame: From first dose up to 30 days post last dose. (an average of 50.3 weeks up to a maximum of 128 weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
Participants
  All grade | 38
  Grade 3/4 | 30

3. Secondary Outcome: Number of Participants and Severity of Treatment Related All Grade Adverse Events (AEs) and Grade 3/4 AEs
Description: Number of participants and severity of treatment related all grade adverse events (AEs) and grade 3/4 AEs as per NCI CTCAE.
Time Frame: From first dose up to 30 days post last dose. (an average of 50.3 weeks up to a maximum of 124 weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
Participants
  All grade | 34
  Grade 3/4 | 13

4. Secondary Outcome: Mean Change From Baseline in Hematology Laboratory Analysis - Hemoglobin
Description: Mean change from baseline in hematology laboratory analysis - hemoglobin
Time Frame: at Cycle 4 Day 1 and Cycle 7 Day 1
Population: all treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
g/dL
  cycle 4 day 1: number analyzed (Participants) | 30
  cycle 4 day 1 | -1.16 (1.431)
  cycle 7 day 1: number analyzed (Participants) | 21
  cycle 7 day 1 | -1.13 (1.127)

5. Secondary Outcome: Mean Change From Baseline in Hematology Laboratory Analysis - Erythrocytes
Description: Mean change from baseline in hematology laboratory analysis - erythrocytes.
  Baseline value is defined as the last value or measurement taken prior to the first dose in the study
Time Frame: at Cycle 4 Day 1 and Cycle 7 Day 1
Population: all treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: 10¹²Cells/L
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
10¹²Cells/L
  cycle 4 day 1: number analyzed (Participants) | 30
  cycle 4 day 1 | -0.60 (0.567)
  cycle 7 day 1: number analyzed (Participants) | 21
  cycle 7 day 1 | -0.67 (0.609)

6. Secondary Outcome: Mean Change From Baseline in Hematology Laboratory Analysis - Platelets, Leukocytes and Neutrophils
Description: Mean change from baseline in hematology laboratory analysis - platelets, leukocytes and neutrophils.
  Baseline value is defined as the last value or measurement taken prior to the first dose in the study
Time Frame: at Cycle 4 Day 1 and Cycle 7 Day 1
Population: all treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: 10⁹Cells/L
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
10⁹Cells/L
  Baseline Platelets: number analyzed (Participants) | 37
  Baseline Platelets | 0 (0)
  cycle 4 day 1 - platelets: number analyzed (Participants) | 29
  cycle 4 day 1 - platelets | 13.8 (135.86)
  cycle 7 day 1 - platelets: number analyzed (Participants) | 20
  cycle 7 day 1 - platelets | 11.7 (131.25)
  cycle 4 day 1 - leukocytes: number analyzed (Participants) | 30
  cycle 4 day 1 - leukocytes | -15.481 (21.6350)
  cycle 7 day 1 - leukocytes: number analyzed (Participants) | 21
  cycle 7 day 1 - leukocytes | -15.127 (18.5744)
  cycle 4 day 1 - neutrophils: number analyzed (Participants) | 30
  cycle 4 day 1 - neutrophils | -10.064 (14.2661)
  cycle 7 day 1 - neutrophils: number analyzed (Participants) | 21
  cycle 7 day 1 - neutrophils | -10.495 (13.5489)

7. Secondary Outcome: Mean Change From Baseline in the Percentage of Blasts/Leukocytes in Hematology Laboratory Analysis
Description: Mean change from baseline in hematology laboratory analysis - blasts/leukocytes
  Baseline value is defined as the last value or measurement taken prior to the first dose in the study
Time Frame: at Cycle 4 Day 1 and Cycle 7 Day 1
Population: all treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: Percentage of blasts/leukocytes
Arm/Group | Fedratimib
Number analyzed (Participants) | 31
Percentage of blasts/leukocytes
  cycle 4 day 1: number analyzed (Participants) | 22
  cycle 4 day 1 | 0.0 (1.50)
  cycle 7 day 1: number analyzed (Participants) | 15
  cycle 7 day 1 | -0.2 (1.82)

8. Secondary Outcome: Mean Change From Baseline in Chemistry Parameters Analysis - ALT, AST, Amylase, Lipase
Description: Mean change from baseline in chemistry parameters analysis - ALT, AST, Amylase, Lipase
  Baseline value is defined as the last value or measurement taken prior to the first dose in the study
Time Frame: at Cycle 4 Day 1 and Cycle 7 Day 1
Population: all treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
U/L
  cycle 4 day 1 - ALT: number analyzed (Participants) | 33
  cycle 4 day 1 - ALT | 0.7 (18.49)
  cycle 7 day 1 - ALT: number analyzed (Participants) | 23
  cycle 7 day 1 - ALT | 7.3 (29.53)
  cycle 4 day 1 - AST: number analyzed (Participants) | 33
  cycle 4 day 1 - AST | -0.9 (8.71)
  cycle 7 day 1 - AST: number analyzed (Participants) | 23
  cycle 7 day 1 - AST | 2.3 (11.83)
  cycle 4 day 1 - Amylase: number analyzed (Participants) | 33
  cycle 4 day 1 - Amylase | 15.1 (17.17)
  cycle 7 day 1 - Amylase: number analyzed (Participants) | 23
  cycle 7 day 1 - Amylase | 10.5 (15.19)
  cycle 4 day 1 - Lipase: number analyzed (Participants) | 33
  cycle 4 day 1 - Lipase | 11.6 (19.22)
  cycle 7 day 1 - Lipase: number analyzed (Participants) | 23
  cycle 7 day 1 - Lipase | 6.4 (13.60)

9. Secondary Outcome: Mean Change From Baseline in Chemistry Parameters Analysis - Creatinine
Description: Mean change from baseline in chemistry parameters analysis - Creatinine.
  Baseline value is defined as the last value or measurement taken prior to the first dose in the study
Time Frame: at Cycle 4 Day 1 and Cycle 7 Day 1
Population: all treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
umol/L
  cycle 4 day 1 - Creatinine: number analyzed (Participants) | 33
  cycle 4 day 1 - Creatinine | 23.9 (18.82)
  cycle 7 day 1 - Creatinine: number analyzed (Participants) | 23
  cycle 7 day 1 - Creatinine | 28.5 (23.03)

10. Secondary Outcome: Spleen Response Rate by Palpation
Description: Spleen response rate by palpation is the percentage of participants with a spleen response according to the IWG-MRT 2013 at the end of Cycle 6 as compared to baseline. This will be calculated for participants that have an enlarged spleen (≥ 5 cm below LCM) at baseline. Participants with a missing spleen size assessment at the end of Cycle 6 including those who meet the criteria for progression of splenomegaly before the end of Cycle 6 will be considered not to be responders.
Time Frame: From First Dose to end of Cycle 6 (approximately 168 days)
Population: Palpation evaluable population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 37
Percentage of Participants | 16.2 [6.2 to 32.0]

11. Secondary Outcome: Symptom Response Rate
Description: Symptom response rate (SRR) is defined as the percentage of participants with ≥ 50% reduction from baseline to the end of Cycle 6 in total symptom score (TSS) measured by MFSAF version 4.0. The TSS will be defined as the sum of each of the 7 symptom scores. Participants without a baseline TSS > 0 will be considered non-evaluable (due to no place for symptom reduction) for the SRR analysis. Participants with a missing TSS at the end of Cycle 6 or who had disease progression before the end of the Cycle 6 will be considered non-responders.
Time Frame: From First Dose to end of Cycle 6 (approximately 168 days)
Population: MFSAF Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 36
Percentage of participants | 44.4 [27.9 to 61.9]

12. Secondary Outcome: Durability of Spleen Volume Response by MRI/CT (DR)
Description: Durability of spleen volume response (DR) by MRI/CT is defined as time from the first documented spleen response (ie, ≥ 35% reduction in spleen volume) to the date of subsequent progressive disease (PD) (ie, ≥ 25% increase in spleen volume from baseline) or death, whichever is earlier. In the absence an event (ie, subsequent spleen volume reduction < 35% before the analysis is performed), the DR will be censored at the date of the last valid assessment performed before the analysis performed date. Durability of spleen volume response by MRI/CT scan will be analyzed using Kaplan-Meier method.
Time Frame: From Cycle 1 Day 1 up to 30 days after last dose (Approximately an average of 59.40 Weeks)
Population: EE population, Responders only
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Fedratimib
Number analyzed (Participants) | 24
Weeks | 115.1 [38.1 to NA] — ULN not reached. 15 participants were censored. Insufficient number of events (subsequent progressive disease or deaths) occurred to calculate the ULN via the K-M method.

13. Secondary Outcome: Durability of Spleen Response by Palpation (DRP)
Description: Durability of spleen response by palpation (DRP) is defined as time from the date of first documented palpable spleen response, according to the IWG-MRT 2013 to the date of subsequent PD according to the IWG-MRT 2013 or death, whichever is earlier. Durability of spleen response by palpation according to the IWG-MRT 2013 criteria will be calculated for subjects that have an enlarged spleen at baseline (≥ 5 cm below LCM), and that have a spleen response by palpation. In the absence of an event (ie, no loss of spleen response by palpation) before the analysis is performed, the DRP will be censored at the date of the last valid assessment performed before the analysis performed date. Durability of spleen response by palpation will be analyzed using Kaplan-Meier (K-M) method.
Time Frame: From Cycle 1 Day 1 up to 30 days after last dose (Approximately an average of 59.32 Weeks)
Population: Palpation Evaluable Population, responders only
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Fedratimib
Number analyzed (Participants) | 21
Weeks | 134.9 [33.3 to NA] — ULN not reached. 14 participants were censored. Insufficient number of events (subsequent progressive disease or deaths) occurred to calculate the ULN via the K-M method.

14. Secondary Outcome: Durability of Symptom Response (DSR)
Description: Durability of symptoms response is defined as time from the first documented response in TSS (ie, reduction in TSS ≥ 50%) measured by MFSAF version 4.0 to the first documented TSS reduction < 50%. In the absence of TSS reduction < 50% before the analysis performed, the DSR will be censored at the date of the last valid assessment performed before the analysis performed date.
Time Frame: From Cycle 1 Day 1 up to 30 days after last dose (Approximately an average of 31.33 Weeks)
Population: MFSAF population, Responders only
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Fedratimib
Number analyzed (Participants) | 28
Weeks | 20.1 [11.0 to 48.0]

15. Secondary Outcome: Number of Participants With Grade 3 or Higher AEs: Nausea, Vomiting, Diarrhea and Encephalopathy Including Wernicke's.
Description: Number of participants with grade 3 or higher AEs: Nausea, Vomiting, Diarrhea and Encephalopathy including Wernicke's.
Time Frame: From first dose to end of treatment (an average of 50.3 weeks up to a maximum of 124 weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
Participants
  Nausea: number analyzed (Participants) | 12
  Nausea | 0
  Vomitting: number analyzed (Participants) | 12
  Vomitting | 0
  Diarrhea: number analyzed (Participants) | 12
  Diarrhea | 0
  Encephalopathy | 0
  Wernickes Encephalopathy | 0

16. Secondary Outcome: Number of Participants With Thiamine Levels < Lower Limit of Normal (LLN).
Description: Number of participants with thiamine levels < LLN.
  LLN of thiamine is 70 nmol/L.
Time Frame: At Cycle 1, 2, 3, and every 3 cycles afterwards till End of Treatment (an average of 50.3 weeks up to a maximum of 124 weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
Participants
  Cycle 1: number analyzed (Participants) | 37
  Cycle 1 | 0
  Cycle 2: number analyzed (Participants) | 31
  Cycle 2 | 2
  Cycle 3: number analyzed (Participants) | 30
  Cycle 3 | 2
  Cycle 6: number analyzed (Participants) | 23
  Cycle 6 | 0
  Cycle 9: number analyzed (Participants) | 15
  Cycle 9 | 0
  Cycle 12: number analyzed (Participants) | 10
  Cycle 12 | 0
  Cycle 15: number analyzed (Participants) | 13
  Cycle 15 | 0
  Cycle 18: number analyzed (Participants) | 12
  Cycle 18 | 0
  Cycle 21: number analyzed (Participants) | 10
  Cycle 21 | 0
  Cycle 24: number analyzed (Participants) | 8
  Cycle 24 | 0
  Cycle 27: number analyzed (Participants) | 8
  Cycle 27 | 0
  Cycle 30: number analyzed (Participants) | 5
  Cycle 30 | 0
  Cycle 33: number analyzed (Participants) | 4
  Cycle 33 | 0
  Cycle 36: number analyzed (Participants) | 4
  Cycle 36 | 0
  Cycle 39: number analyzed (Participants) | 6
  Cycle 39 | 0
  Cycle 42: number analyzed (Participants) | 5
  Cycle 42 | 0
  Cycle 45: number analyzed (Participants) | 3
  Cycle 45 | 0
  Cycle 48: number analyzed (Participants) | 4
  Cycle 48 | 0
  Cycle 51: number analyzed (Participants) | 2
  Cycle 51 | 0
  cycle 54: number analyzed (Participants) | 1
  cycle 54 | 0
  End of Treatment: number analyzed (Participants) | 20
  End of Treatment | 1
  Total number of participants with thiamine <LLN | 5

17. Secondary Outcome: Number of Participants With Thiamine Levels > Upper Limit of Normal (ULN).
Description: Number of participants with thiamine levels > ULN.
  ULN of thiamine is 180 nmol/L.
Time Frame: as for outcome 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
Participants
  Cycle 1: number analyzed (Participants) | 37
  Cycle 1 | 21
  Cycle 2: number analyzed (Participants) | 31
  Cycle 2 | 9
  Cycle 3: number analyzed (Participants) | 30
  Cycle 3 | 9
  Cycle 6: number analyzed (Participants) | 23
  Cycle 6 | 6
  Cycle 9: number analyzed (Participants) | 15
  Cycle 9 | 5
  Cycle 12: number analyzed (Participants) | 10
  Cycle 12 | 4
  Cycle 15: number analyzed (Participants) | 13
  Cycle 15 | 7
  Cycle 18: number analyzed (Participants) | 12
  Cycle 18 | 4
  Cycle 21: number analyzed (Participants) | 10
  Cycle 21 | 4
  Cycle 24: number analyzed (Participants) | 8
  Cycle 24 | 3
  Cycle 27: number analyzed (Participants) | 8
  Cycle 27 | 2
  Cycle 30: number analyzed (Participants) | 5
  Cycle 30 | 2
  Cycle 33: number analyzed (Participants) | 4
  Cycle 33 | 2
  Cycle 36: number analyzed (Participants) | 4
  Cycle 36 | 0
  Cycle 39: number analyzed (Participants) | 6
  Cycle 39 | 2
  Cycle 42: number analyzed (Participants) | 5
  Cycle 42 | 1
  Cycle 45: number analyzed (Participants) | 3
  Cycle 45 | 1
  Cycle 48: number analyzed (Participants) | 4
  Cycle 48 | 3
  Cycle 51: number analyzed (Participants) | 2
  Cycle 51 | 1
  Cycle 54: number analyzed (Participants) | 1
  Cycle 54 | 0
  End of Treatment: number analyzed (Participants) | 20
  End of Treatment | 9
  Total number of participants with thiamine > ULN | 28

18. Secondary Outcome: Number of Participants With Clinically Notable Laboratory Results, Grade 3 or 4
Description: Number of participants with clinically notable laboratory results, Grade 3 or 4
Time Frame: From first dose up to 30 days post last dose. (an average of 50.3 weeks up to a maximum of 124 weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratimib
Number analyzed (Participants) | 38
Participants
  GFR from Creatinine adjusted for BSA (mL/min/1.73m²) | 7
  Gamma Glytamyl Transferase (U/L) | 2
  Lipase (U/L) | 2
  Potassium (mmol/L): number analyzed (Participants) | 37
  Potassium (mmol/L) | 1
  Sodium (mmol/L) | 4
  Triglycerides (mmol/L): number analyzed (Participants) | 22
  Triglycerides (mmol/L) | 1
  Hemoglobin (g/dL) | 20
  Leukocytes (10⁹/L) | 5
  Lymphocytes (10⁹/L) | 7
  Neutrophils, Segmented (10⁹/L) | 4
  Neutrophils, Segmented and Band Form (10⁹/L) | 2
  Platelets (10⁹/L) | 10
  Prothrombin INR (ratio): number analyzed (Participants) | 27
  Prothrombin INR (ratio) | 1

ADVERSE EVENTS:
Time Frame: Adverse Events: From first dose up to 30 days post last dose. (An average of 50.3 weeks up to a maximum of 124 weeks) All-Cause Mortality: From first dose up to LPLV PE final Database lock: approximately 56 Months.
Description: Adverse events will be analyzed in terms of TEAEs that are defined to be any event that begins or worsens in grade after the start of fedratinib through 30 days after the last dose.
Groups:
- Fedratinib: 400 mg/day PO (4 x 100 mg capsules)
Arm/Group | Fedratinib
All-Cause Mortality (participants affected / at risk) | 16/38
Serious Adverse Events (participants affected / at risk) | 22/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fedratinib (N=38)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Cardiac tamponade (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 4
Humerus fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Chronic kidney disease (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fedratinib (N=38)
Anaemia (Blood and lymphatic system disorders) | 23
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Atrial fibrillation (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 2
Lacrimation increased (Eye disorders) | 3
Vision blurred (Eye disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 17
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 16
Stomatitis (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Chills (General disorders) | 4
Early satiety (General disorders) | 2
Fatigue (General disorders) | 12
Influenza like illness (General disorders) | 3
Oedema peripheral (General disorders) | 10
Pain (General disorders) | 3
Peripheral swelling (General disorders) | 4
Pyrexia (General disorders) | 4
Bacteraemia (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 2
Candida infection (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 5
Contusion (Injury, poisoning and procedural complications) | 7
Fall (Injury, poisoning and procedural complications) | 5
Skin laceration (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 3
Amylase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blast cell count increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 14
Glomerular filtration rate decreased (Investigations) | 4
Lipase increased (Investigations) | 3
Vitamin B1 decreased (Investigations) | 7
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 9
Gout (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Disturbance in attention (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 10
Encephalopathy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 9
Acute kidney injury (Renal and urinary disorders) | 4
Dysuria (Renal and urinary disorders) | 3
Pollakiuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 3
Onychoclasis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 10
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03755518/Prot_SAP_000.pdf